CLINICAL TRIAL: NCT07141953
Title: The Effect of Yoga on Quality of Life, Sleep Quality, and Spiritual Well-Being in Women Who Undergo Surgical Menopause Following Gynecological Cancer Surgery: A Randomized Controlled Trial
Brief Title: Yoga in Women With Surgical Menopause After Gynecological Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Selcan Zeynep Ergöz Aksoy, RN. MSc., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DEU-2025/12-14
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Gynecological Oncology; Gynecology; Oncology; Surgical Menopause; Symptom Management; Quality of Life; Sleep Quality; Well-being; Yoga; Yoga for Cancer
Keywords: gynecological oncology; gynecology; oncology; surgical menopause; symptom management; quality of life; sleep quality; well-being; yoga; yoga for cancer
MeSH Terms: conditions — Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Yoga

STUDY DESIGN:
Intervention Model Description: This study was designed as a prospective and Randomized Controlled experimental study. Participants were randomly divided into two groups in a 1:1 ratio; the study group and the control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Individuals who perform yoga
  Interventions: Behavioral: Yoga
- Control Group (No Intervention): Controls

INTERVENTIONS:
Behavioral: Yoga — Participants in the intervention group will take part in an 8-week yoga program designed for women who have entered surgical menopause after gynecological cancer surgery. The program will consist of two 60-minute sessions per week, one delivered online and one delivered face-to-face, conducted in small groups (5-6 participants) or individually, depending on participant availability. The sessions will include physical postures, breathing exercises, and relaxation/meditation techniques. The program will be delivered by a certified yoga instructor.
  Arms: Study Group

SUMMARY:
This randomized controlled trial investigates the effects of yoga on quality of life, sleep quality, and spiritual well-being in women who have entered surgical menopause after gynecological cancer surgery. Yoga is expected to be a supportive intervention for symptom management and to improve overall well-being in this patient population.

DETAILED DESCRIPTION:
Surgical menopause after gynecological cancer surgery is associated with sudden and severe symptoms that may reduce quality of life, disturb sleep, and affect overall well-being. Supportive non-pharmacological approaches such as yoga may help manage these challenges.

This randomized controlled trial will investigate the effects of an 8-week yoga program on quality of life, sleep quality, and spiritual well-being in women who have entered surgical menopause. Forty-six participants will be randomly assigned to either a yoga intervention group or a control group. The intervention group will attend two yoga sessions per week (one online, one face-to-face) in small groups or individually with a certified instructor, while the control group will receive usual care and be offered yoga after the study.

Assessments will be conducted at baseline, post-intervention (8 weeks), and 3-month follow-up using standardized questionnaires. It is expected that yoga will support symptom management and improve overall well-being in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Age between 18-65 years Diagnosis of primary gynecological cancer (ovarian, endometrial, cervical, vaginal, or vulvar) (Stage I-III) Ability to read, understand, and speak Turkish Completion of all adjuvant treatments (surgery, chemotherapy, and/or radiotherapy) at least 6 months prior Access to the internet Having a computer/tablet/phone with a camera Willingness and ability to attend at least 80% of the yoga sessions Voluntary participation in the study

Exclusion Criteria:

Any condition that prevents communication Cognitive, sensory, or physical impairment that prevents yoga practice Diagnosis of metastatic gynecological cancer Regular yoga practice within the last 6 months (at least once a week for 8 consecutive weeks)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life with yoga | Baseline, 2 months (end of intervention), and 5 months (3-month follow-up)
  Change in WHOQOL-BREF total score. Scores range 0-100; higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Change in Sleep Quality | Baseline, 2 months (end of intervention), and 5 months (3-month follow-up)
  Change in Pittsburgh Sleep Quality Index (PSQI). Higher scores indicate worse sleep quality.
Change in Spiritual Well-Being | Baseline, 2 months (end of intervention), and 5 months (3-month follow-up)
  Change in FACIT-Sp-12 total score. Higher scores indicate greater spiritual well-being.
Change in Menopausal Symptoms | Baseline, 2 months (end of intervention), and 5 months (3-month follow-up)
  Change in Menopause Rating Scale total score. Higher scores indicate greater symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Bilgiç, Prof., Study Director — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Balçova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33127864/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19214594/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23387909/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29452777/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25739642/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25845383/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27261993/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32168205/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30168358/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22502670/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12008794/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32059825/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35191141/